CLINICAL TRIAL: NCT07266194
Title: A Double-Blind Observational Study to Validate the SpotitEarly Test for the Detection of Breast Cancer
Brief Title: The Study Will Enroll Females Who Are Coming in for Their Annual Mammogram Screening and Who Are Schedule for a Biopsy to Provide a Breath Sample Via a Mask to Evaluate if Breast Cancer Can be Detected.
Status: Not yet recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: SpotitEarly (Industry)
Responsible Party: Principal Investigator, Brian Englander, Chair of Department of Radiology at Pennsylvania Hospital, Abramson Cancer Center at Penn Medicine
Other Study IDs: 859242
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Detection
Keywords: Breast cancer; Screening; Breath Samples; Cancer Detection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Target Population Arm: Women scheduled for routine breast cancer screening.
  Interventions: Other: Breathing Mask
- Enriched Arm: Women scheduled for breast biopsy with a Breast Imaging and Reporting Data System (BI-RADS®) score of 4B or above
  Interventions: Other: Breathing Mask

INTERVENTIONS:
Other: Breathing Mask — Breath sample collection using a sample collection kit

SUMMARY:
Primary Objective:

1. To evaluate the sensitivity of the SpotitEarly test for breast cancer detection in women

Secondary Objectives:

1. To evaluate the performance of the SpotitEarly in various subgroups.
2. To evaluate the performance of the SpotitEarly test in detecting early-stage cancer (stages 0-2).
3. To assess whether the performance of the SpotitEarly test is affected by psychological impacts (e.g. anxiety) related to the biopsy procedure.

Exploratory Objective:

1. To evaluate the test-retest reliability of SpotitEarly's test.

DETAILED DESCRIPTION:
The goal of this study is to find out whether a system that uses trained detection dogs and artificial intelligence (AI) can identify breast cancer from a person's breath. Women who are scheduled to have screening breast cancer screening, or a biopsy for a possible cancer, will be invited to take part. Participants will be asked to breathe into a surgical mask to collect a breath sample.

The mask will be sent to a special laboratory, where trained dogs and an AI-based system will check the sample for signs of breast cancer. The results from the dogs and AI will be compared to the actual results from the medical screening or biopsy to see how accurate the system is at detecting breast cancer.

ELIGIBILITY:
Inclusion Criteria for Arm 1 (Target Population Arm)

1. 40 years of age and above. OR Between 18 and 39 years of age (inclusive) and a carrier of germline pathogenic variants associated with high risk of breast cancer: BRCA1, BRCA 2, PTEN, TP53, CDH1 or STK11 OR Between 18 and 39 years of age (inclusive) with a family history of breast or ovarian cancer involving at least one first or two second-degree relatives who were diagnosed with breast or ovarian cancer before the age of 50 years.
2. Assign female at birth.
3. Scheduled for routine annual breast cancer screening
4. Capable of giving consent for self, which includes compliance with the requirements and restriction listed in the Informed Consent and in the protocol.

Inclusion Criteria for Arm 2 (Enriched Arm)

1. 40 years of age and above. OR Between 18 and 39 years of age (inclusive) and a carrier of germline pathogenic variants associated with high risk of breast cancer: BRCA1, BRCA 2, PTEN, TP53, CDH1 or STK11 OR Between 18 and 39 years of age (inclusive) with a family history of breast or ovarian cancer involving at least one first or two second-degree relatives who were diagnosed with breast or ovarian cancer before the age of 50 years.
2. Assigned female at birth
3. Scheduled for breast biopsy.
4. BI-RADS® screening score of 4B or above
5. Capable of giving consent for self, which includes compliance with the requirements and restriction listed in the Informed Consent and in the protocol.

Exclusion Criteria (Both Arms)

1. Diagnosis with cancer within the past year. Individuals who underwent surgical removal of cancerous non-metastatic skin lesions can be recruited.
2. Has received any cancer treatments within the past year.
3. Has participated in another clinical study within the last 30 days.
4. Had bilateral surgery for breast cancer or for preventive reasons related to breast cancer.
5. Had a medical procedure in the chest cavity and/or airways within the past 2 weeks, which may interfere with the ability to provide a normal breath sample as required by the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible subjects who are seen at Pennsylvania Hospital for their breast cancer screening and biopsy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specifically of the SpotitEarly testing in each of the subgroups | 12 months
  Age: under 40, 40-49, 50-64, 65 and older. Race: White, Black/African American, Asian and Pacific Islander, Native American/ Alaska Native, more than one race.
  Germline pathogenic variant carriers associated with high risk for breast cancer (BRCA1, BRCA2, PTEN, TP53, CDH1, STK11) versus non-carriers.
  Smoking status: smokers versus non-smokers. Women with type-2 diabetes versus women who were not diagnosed with the disease.

SECONDARY OUTCOMES:
Sensitivity of the SpotitEarly test in detecting early-stage cancer among breast cancer-positive samples | 24 months
  he test's specificity and its confidence interval (CI) will be analyzed in the following subgroups: Negative non-benign samples in Arm 1. All benign samples in Arm 1. Benign samples in Arm 1 of participants with a BI-RADS® score of 4B or above. Benign samples in Arm 2.

CONTACTS AND LOCATIONS:
Overall Officials: Brian S Englander, MD, Principal Investigator — Penn Medicine; Brian S. Englander, MD, Principal Investigator — Penn Medicine